CLINICAL TRIAL: NCT00154973
Title: Expression of Hypoxia-Inducible Factor-α in Oral Precancers and Cancers
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9261701447
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2005-09-12 (Estimated); Status verified 2004-08

CONDITIONS: Oral Cancer
Keywords: oral precancers; oral cancer; hypoxia-inducible factor
MeSH Terms: conditions — Mouth Neoplasms

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
Expression of hypoxia-inducible factor-α in oral precancers and cancers

DETAILED DESCRIPTION:
Expression of hypoxia-inducible factor-α in oral precancers and cancers

ELIGIBILITY:
Inclusion Criteria:

* oral cancer specimens

Exclusion Criteria:

* not oral cancer specimens

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2004-08; Study Completion 2005-06

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Pin Chiang, DMSc, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan